CLINICAL TRIAL: NCT02513173
Title: Effects of Different Verbal Instructions on Lumbar Multifidus Muscle Activation in Healthy and Patients With Low Back Pain
Brief Title: Effects of Different Verbal Instructions in Healthy Adults and Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Other Study IDs: TWU17581
Record Dates: First submitted 2015-07-24; First posted 2015-07-31 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2015-07

CONDITIONS: Low Back Pain
Keywords: low back pain; verbal instruction; lumbar multifidus; ultrasound imaging; Muscle thickness
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low back pain group: No intervention
- Control: No intervention

SUMMARY:
Segmental stabilization exercise has been shown to be effective in the rehabilitation of low back pain (LBP). Due to the isometric nature of segmental stabilization exercise, manual therapists use various verbal instructions to elicit lumbar multifidus muscle contraction. The purpose of this study was to assess whether or not three verbal instructions would alter muscle thickness of the lumbar multifidus differently in asymptomatic individuals and patients with LBP.

Three verbal instructions were selected for this study: (1) swell the muscle underneath the transducer, (2) draw your belly button in towards your spinal column, and (3) think about tilting your pelvis but without really doing it. Lumbar multifidus muscle thickness was determined using parasagittal ultrasound imaging. Measurements of muscle thickness were collected at rest and during verbal instructions from 21 asymptomatic adults and 21 patients with LBP. Percent changes of muscle thickness during contraction and at rest were compared between groups and across verbal instructions.

DETAILED DESCRIPTION:
Participants:

Eligible participants were English-speaking adults 18 years of age or older. Additional criteria for asymptomatic healthy adults included no existing low back pain (LBP) and no LBP in the past year. Additional criteria for patient participants included existing LBP near the L5-S1 level with an average pain intensity score ≥ 2/10 (numeric pain rating scale of 0-10, 0 being no pain, 10 being unbearable pain).

Exclusion criteria for all participants included previous low back surgery, systemic joint disease (e.g. rheumatoid arthritis), cancer of the lower quadrant, neurological disorders, allergic reaction to ultrasound gel, or inability to obtain testing positions (prone lying).

After participants were informed of the risks, benefits and procedures of the study, they were asked to sign a written consent form approved by the TWU Institutional Review Board - Dallas. Eligible participants were asked to complete an intake form, asking them about their age, gender, and past medical history. For participants with existing LBP, they were asked about their pain location, duration, intensity, and nature of their existing LBP and their LBP history. The height and body weight of each participant were taken to determine the body mass index (BMI). BMI has been shown to be a factor affecting muscle size.

Instrumentation:

1. The Modified Oswestry Low Back Pain Index (OSW) questionnaire was used to determine an individual's perceived disability and function limitation due to his/her low back pain. The OSW questionnaire has been shown to be reliable and valid.
2. A Sonosite M-Turbo ultrasound scanner (Sonosite, Inc., Bothell, WA) was used to measure muscle size of the lumbar multifidus. A curvilinear transducer (3-5 MHz) will be used to take transverse images of segmental lumbar multifidus at the L5-S1 segment. If the patient has multiple painful segments, the most painful segment will be imaged. The most common painful segments are L4-5 or L5-S1 in patients with LBP.
3. The ImageJ software (free download from the NIH website) was used to determine muscle thickness off-line.

US Image Acquisition:

Participants was lying in prone on an examination table with their arms on the sides. A pillow was placed under the participant's abdomen to flatten the lumbar lordotic curve and an inclinometer was placed on the lumbosacral junction to ensure the lumbar curve ≤10.

The right side of asymptomatic healthy adults and the painful side of patients with low back pain were imaged. The spinous processes of the right L5-S1 or the painful segment were identified by palpation and marked with an erasable pen. Next, the spinous process was verified using US imaging. Transverse images of the segmental multifidus muscle were captured by placing the transducer horizontally on the spinous process of the target segment. The transverse image of segmental lumbar multifidus was taken 3 times "at rest" and 3 times during muscle activations of the lumbar multifidus. Activation of lumbar multifidus was achieved by asking participants to generate a slow gentle sustained (isometric) contraction of the lumbar multifidus using 3 different verbal instructions without moving their spine or pelvis. Participants held each contraction for 3-5 seconds. The order of 3 verbal instructions was given in a random order to minimize the learning and fatigue effects. Therefore, each participant performed a total of 9 lumbar multifidus muscle contractions during each testing session. Prior to taking ultrasound images, the anatomy and location of the lumbar multifidus muscle were explained and shown to participants using a model and pictures. Next, the following 3 verbal instructions were used to generate a multifidus contraction:

Breathe in and out and:

1. Without moving your spine, try to "swell" the muscle underneath the transducer.
2. Without moving your spine, draw your spinal column in toward your belly button.
3. Attempt to elongate your spine by drawing the muscles in your back up toward your head.

All participants were asked to return one week later, the procedure was repeated. The order of verbal instructions also was randomized in the 2nd session.

ELIGIBILITY:
Inclusion Criteria:

* additional criteria for asymptomatic healthy adults include no existing LBP and no LBP in the past year.
* additional criteria for patient participants include existing LBP near the L5-S1 level with an average pain intensity score ≥ 2/10 (numeric pain rating scale of 0-10, 0 being no pain, 10 being unbearable pain).

Exclusion Criteria:

* previous low back surgery,
* systemic joint disease (e.g. rheumatoid arthritis),
* cancer of the lower quadrant,
* neurological disorders,
* allergic reaction to ultrasound gel, or
* inability to obtain testing positions (prone lying).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants are English-speaking adults 18 years of age or older, with or without low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic muscle thickness measurement of lumbar multifidus | Participants were measured and then followed-up one week later
  Muscle thickness of lumbar multifidus was measured at rest and during contraction under each of 3 verbal instructions on two visits with an average of one week apart.